CLINICAL TRIAL: NCT04722692
Title: Sentinel Lymph Node Biopsy in Ductal Cancer in Situ or Unclear Lesions of the Breast and How to Not do it. An Open-label, Phase 3, Randomised Controlled Trial. (SentiNot 2.0).
Brief Title: Delayed Sentinel Lymph Node Biopsy in Ductal Cancer in Situ
Acronym: SENTINOT_2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Västmanlands Hospital, Västerås, Sweden (Unknown); Sahlgrenska University Hospital (Other); University Hospital, Linkoeping (Other); Skane University Hospital (Other); Blekinge County Council Hospital (Other); Växjö Hospital, Växjö, Sweden (Unknown); The University of Hong Kong-Shenzhen Hospital (Other); Norrlands University Hospital (Other); Dalarna County Hospital, Falun, Sweden (Unknown); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Andreas Karakatsanis, Principal Investigator, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UUBreast01
Record Dates: First submitted 2020-12-23; First posted 2021-01-25 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: DCIS; Breast Cancer; Breast Neoplasms; Sentinel Lymph Node
Keywords: Sentinel Lymph Node Dissection; DCIS; Ductal Cancer In situ of the breast; Breast cancer; Superparamagnetic Iron Oxide Nanoparticles; Sentinel Lymph Node; Risk reducing mastectomy
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will have been injected with SPIO during the breast procedure. Those who have invasive breast cancer on final pathology will receive radioisotope and undergo SLND. Patients will be randomly allocated to one of two arms: Experimental arm (SLND will be SPIO-guided and the isotope activity will be controlled as background) and control arm (SLND will be isotope-guided and SPIO activity will be controlled as background).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delayed SLND (SPIO-first arm) (Experimental): All study participants have been injected interstitially with SPIO, 2ml, at the primary operation. Magnetic axillary signal is registered at the end of the procedure but the SLN is not removed. If invasive cancer is found in the specimen, reoperation for SLND with the addition of Tc +/- BD is performed.
  At reoperation, SPIO is the "primary" detection tracer.
  Interventions: Diagnostic Test: Delayed SLND
- Late SLND (RI-first arm) (Active Comparator): All study participants have been injected interstitially with SPIO, 2ml, at the primary operation. Magnetic axillary signal is registered at the end of the procedure but the SLN is not removed. If invasive cancer is found in the specimen, reoperation for SLND with the addition of Tc +/- BD is performed.
  At reoperation, Tc is the "primary" detection tracer.
  Interventions: Diagnostic Test: Late SLND

INTERVENTIONS:
Diagnostic Test: Delayed SLND — SLND performed after surgery for DCIS or other pre-invasive lesions, where final pathology showed invasive breast cancer. Patients have received SPIO in the breast at the first operation, prior to dissection and resection and the SLN has already been marked with SPIO. These SLNs are to be removed.
  SLND is divided into the following steps:
  1. Transcutaneous signal
  2. Incision in the axilla (skin, subcutaneous fat and fascia) and "In situ" signal
  3. SLN identification "in situ"
  4. SLN excision and signal "ex vivo"
  5. Background axillary counts. For step "d" the radioactive counts are registered for each SLN that has been excised. When the procedure is completed successfully with SPIO, then background axillary isotope counts are registered and, if present, SLND continues as described above with the isotope as primary tracer.
  Arms: Delayed SLND (SPIO-first arm)
Diagnostic Test: Late SLND — SLND performed after surgery for DCIS or other pre-invasive lesions, where final pathology showed invasive breast cancer. Patients will be injected with radioisotope in the operated breast before SLND according to standard of care. Any SLNs detected with this intervention are to be removed.
  SLND is divided into the following steps:
  1. Transcutaneous signal
  2. Incision in the axilla (skin, subcutaneous fat and fascia) and "In situ" signal
  3. SLN identification "in situ"
  4. SLN excision and signal "ex vivo"
  5. Background axillary counts. For step "d" the magnetic counts are registered for each SLN that has been excised. When the procedure is completed successfully with the isotope, then background axillary iSPIO counts are registered and, if present, SLND continues as described above with the SPIO as primary tracer.
  Arms: Late SLND (RI-first arm)

SUMMARY:
The trial aims to investigate the use of superparamagnetic iron oxide (SPIO) nanoparticles as a tracer for delayed sentinel lymph node dissection (d-SLND) in patients where upfront axillary surgery (SLND) is oncologically deemed unnecessary and should be avoided. This includes but is not limited to patients with a preoperative diagnosis of ductal cancer in situ of the breast (DCIS), an unclear BIRADS 4-5 planned for diagnostic excision or women planned for risk reducing mastectomy. SPIO is injected in the primary operation, and should final specimen pathology demonstrate invasive breast cancer, only then is an operation in the axilla (d-SLND) performed.

DETAILED DESCRIPTION:
The SentiNot 2.0 protocol aims to elucidate the effectivity and accuracy of the delayed sentinel lymph node dissection concept (dSLND) when upfront SLND is considered unnecessary, such as in the setting of a preoperative diagnosis of DCIS, in cases of unclear BIRADS 4 or 5 lesions that are planned for diagnostic excisional biopsy or in selected cases of risk reducing mastectomy. Acknowledging the large variance of practice in this setting, the study aims to address pragmatism to allow for inclusion. For this reason, the trial is designed separately and independently for mastectomy and breast conserving surgery, so that participating sites can recruit as fitting in their practice.

In patients included in the SentiNot 2.0 trial, SPIO (MagTrace,2.0 ml) is injected up to 24 hours preoperatively or perioperatively during primary breast surgery on patients with a preoperative diagnosis of DCIS (or suspicious lesions with no clear diagnosis of invasive cancer but, considered for SLND). The SPIO is injected close to the lesion. If injected less than 24 hours before the operation, a 5 minute massage should be performed. Planned breast surgery is performed. The transcutaneous magnetic counts by SentiMag in the axilla is measured at the end of the breast procedure, so as to allow for confirmation that SLND may be identified. Thus,the SLN is consequently marked with SPIO, but not excised.

In this manner, women that have pure DCIS on final histopathological examination have avoided unnecessary upfront SLND.

If there is underlying invasive breast cancer on final histopathological examination, SLND will be performed at a second operation (d-SLND). A preoperative injection of radioisotope (RI) RI will be added to maximize the chance to detect the SLN. SLND will start with a registration of the magnetic and isotope signal in the axilla, and the incision will be placed in relation to the signal. In patients that have undergone mastectomy, tracers are to be injected intracutaneously in the lateral part of the mastectomy scar. The routine use of blue dye (BD) is strongly advised, but is not compulsory. However, if no transcutaneous signal for SPIO and RI is measured in the axilla pre-incision, an injection of BD according local routines will be administered. Subsequently, SLND will be performed. Patients with upgrade to invasive cancer will undergo SLND, but will be randomized with an allocation ratio of 1:1 to SentiMag first or Radioactive probe first. This will mandate the "principal modality" to perform SLND. Every step of the procedure will be controlled; if the principal modality fails, then the surgeon will use the "secondary". If the principal modality succeeds, the secondary will be registered and documented.

The procedure will be divided to the following steps:

* Transcutaneous axillary signal detection
* Subcutaneous axillary detection, after the incision has been performed.
* In situ SLN identification.
* SLN retrieval ex vivo.
* Residual axillary signal ("Background counts"). If a SLND is successfully completed with the primary modality and no residual axillary signal is detected, before completing the procedure, the secondary modality will be undertaken to allow for the detection of "discordance".

Principle modalities maybe either RI or SPIO. If BD is used, dyed lymphatics should be ignored until failure with both modalities has been reached. The success of each modality, principal and secondary, will be controlled per step. If the surgeon documents principle modality failure for a given step, this is to be documented. The intention-to-treat principle will apply, but if there is failure of the modality randomized as principle, then the per-protocol-analysis principle will apply. All SLNs (magnetic, brown, radioactive, blue) will be removed. Palpable nodes may be removed according to surgeon discretion, but should be reported as such. Total technique failure has to be discussed with the patient in advance, and a plan with patient consent consisting of no-surgery, sampling, axillary dissection or treatment according to intraoperative decision has to be available. If no SLN is found, the procedure performed (axillary clearance, sampling. etc) should be discussed in advance with the patient. The SLN may be sent for frozen section in order to avoid a third operation, if SLN metastases are present.

Standard of care patients (SLND performed upfront for diagnoses included in the inclusion criteria or patients going to l-SLND without SPIO) may also be enrolled in the study prospectively as a control arm.Additionally, patient preference will be tolerated and results will be reported for study secondary and other pre-specified endpoints. Patients in the control group has to be informed that their un-identified data will be used as a comparison and, an oral consent has to be given before surgery regardless whether SLND is planned or not. This will allow for controlled real world data from a prospective control arm in fashion of a cohort.

ELIGIBILITY:
Inclusion Criteria:

A. Preoperative diagnosis of DCIS, of any grade and any size if planned for mastectomy.

B. Planned Risk-reducing mastectomy, if it would be considered for upfront SLND due to institutional practice or in case of an individualised recommendation.

C. Any case with a preoperative diagnosis of pre-invasive or unclear lesion, that upfront SLND would be otherwise considered, such as, but not limited to:

* Patients with a preoperative diagnosis of DCIS grade 3 any size or, DCIS grade 2 larger than or equal to 20 mm on mammography and planned for breast conserving surgery or
* Patients with a preoperative diagnosis of DCIS on core biopsy with a palpable mass on clinical examination or mass effect on radiology or
* Patients with a preoperative diagnosis of DCIS with suspicion of micro-invasion on core biopsy or
* Patients with a mammographic/ultrasound/MRI finding, suspicious for breast cancer (BIRADS 4 or 5) planned for diagnostic excision with breast conserving surgery, with no definitive diagnosis of invasive cancer or
* Patients with a preoperative diagnosis of DCIS, any grade, any size and planned for a complex oncoplastic procedure or
* Patients with a preoperative diagnosis of DCIS, any grade, any size and planned for a procedure that may compromise detection rate for a future SLND, such as, but not confined to: lesions in the upper outer quadrant or the axillary tail, removal of the nipple areola complex and so on or
* The above mentioned categories with a preoperative diagnosis of pleomorphic Lobular Cancer in Situ (pLCIS), classic Lobular Neoplasia (LN) or Atypical Ductal Hyperplasia (ADH).

Exclusion Criteria:

* Intolerance/hypersensitivity to iron, dextran compounds or SPIO
* An iron overload disease
* Patient deprived of liberty or under guardianship
* Pregnant or lactating patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
d-SLND detection rate | One-time (At operation)
  Number of subjects in whom SPIO detected at least one node divided by the number of subjects who underwent the SLND procedure. Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
l-SLND detection rate | One-time (At operation)
  Number of subjects in whom radioisotope detected at least one node divided by the number of subjects who underwent the SLND procedure. Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
Nodal concordance | One-time (At operation)
  Number of nodes identified by both test (SPIO) and control (isotope) out of all nodes identified. Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).

SECONDARY OUTCOMES:
SLND avoidance rate | One-time (At operation)
  Number of subjects with pure DCIS or microinvasive/invasive cancer on specimen pathology who did not undergo SLND out of total number recruited in the trial and injected. Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
Per patient concordance | One-time (At operation)
  Number of subjects in whom at least one node was identified by both test and control out of subjects in whom at least one node was identified by control. Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
Malignancy rate | One-time (At operation)
  Number of subjects in whom at least one malignant lymph node was identified by any method divided by the number of subjects who underwent the SLND procedure. Comparisons and analyses will be performed cumulatively and by type of tracer (SPIO+/-BD vs isotope +/-BD) and per type of surgery (BCT or mastectomy).
Nodal Malignancy rate | One-time (At operation)
  Number of malignant lymph nodes identified by any method divided by the number of nodes who retrieved during SLND procedure. Comparisons and analyses will be performed cumulatively and by type of tracer (SPIO+/-BD vs isotope +/-BD) and per type of surgery (BCT or mastectomy).

OTHER OUTCOMES:
Shoulder Arm Morbidity | Baseline and 1,6,12,24 months postoperatively
  Shoulder Arm Morbidity, assessed by the Disease of the Arm, Shoulder and Hand (DASH) questionnaire. Higher values denote greater disability. Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
Cost effectiveness | Baseline, and at 1, 6 and 12 months postoperatively
  Cost of in-patient and out-patient care, including admission on an out-patient or in-patient basis, operation and anesthesia per minute and SLN pathology, either standard or intraoperative frozen section. Actual expenses will also be registered with respect to costs of admission, anesthesia time, operative time, pathology costs related to axillary procedure (frozen section and routine sectioning), leave of absence, complication related costs and rehabilitation costs. Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
Quality-Adjusted-Life-Years (QALY) | Baseline, and at 1, 6 and 12 months postoperatively
  Incremental cost-effectiveness ratios will be calculated based on the societal costs per Quality-Adjusted-Life-Years (QALY) within 12 months. For calculation of the QALY, the 5-level EQ-5D version (EQ-5D-5L) will be assessed at baseline, and at postoperative visits at 28 days, 6 and 12 months.
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system (5 level Likert items with higher score signifying hiugher problems) and the EQ visual analogue scale (EQ VAS).
Health Related Quality of Life (HR-QoL) | Baseline, and at 1, 6 and 12 months postoperatively
  HR-QoL assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaires core version 30 (EORTC-QLQ-C30). Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
Breast Specific Health Related Quality of Life (HR-QoL) | Baseline, and at 1, 6 and 12 months postoperatively
  HR-QoL assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaires breast version 23 (EORTC-QLQ-B23). Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
Patient reported outcomes and measures | Baseline, and at 1, 6 and 12 months postoperatively
  Patient reported outcomes and measures (PROMS) assessed by the BreastQ questionnaire. Analyses will be performed cumulatively and +/-BD and per type of surgery (BCT or mastectomy).
Disease free interval | 10 years
  Time from operation to local recurrence in the ipsilateral breast either as DCIS or invasive cancer or regional recurrence in the ipsilateral axilla or distant metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Karakatsanis, PhD, Principal Investigator — Uppsala University
Locations (9):
- Baylor College Of Medicine, Houston, Texas, United States
- The University of Hong Kong-Shenzhen Hospital, Hong Kong, Hong Kong
- Sweden (7):
  - Falun Lasarett, Falun, Dalarna County
  - Växjö County Hospital, Vaxjo, Kronoberg County
  - Skåne University Hospital, Lund, Skåne County
  - Västmanland County Hospital, Västerås, Västmanland County
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Uppsala University Hospital, Uppsala
  - Linköping University Hospital, Linköping, Östra Götaland

IPD SHARING:
Plan to Share IPD: No